CLINICAL TRIAL: NCT05481177
Title: Comparative Cohort Study of Post-acute COVID-19 Infection With a Nested, Randomized Controlled Trial of Ivabradine for Those With Postural Orthostatic Tachycardia Syndrome.
Brief Title: Ivabradine for Long-Term Effects of COVID-19 With POTS Cohort
Acronym: COVIVA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Saunders, Colonel, Medical Corps, US Army, Professor of Medicine, Preventive Medicine and Biostatistics, Director, Translational Medicine Unit, Department of Medicine, Director, Division of Clinical Pharmacology and Medical Toxicology, Uniformed Services University of the Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USUHS.2022-094
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Long Haul COVID; Postural Orthostatic Tachycardia Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Postural Orthostatic Tachycardia Syndrome | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Long Haul COVID (No Intervention): Persistent signs and/or symptoms >12 weeks post Covid-infection N = 200 evaluable subjects.
- Post COVID without LHC (No Intervention): No persistent signs and/or symptoms >12 weeks N = 50 evaluable subjects.
- Ivabradine RCT Arms (Placebo Comparator): If POTS or IST is present for participants within either of these cohorts, then they will be assigned to one of two arms of the Ivabradine RCT [2:1 treatment:control].
  RCT Arms: at least 36 evaluable subjects will be enrolled to two arms in a 2:1 ratio. More may be enrolled, depending on the number from the overall COVID-19 cohort who qualify.
  IVA (Ivabradine) - at least 24 evaluable subjects Placebo - at least 12 evaluable subjects
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Ivabradine — Ivabradine is a drug approved to treat tachycardia in volunteers with heart failure. This study is to determine benefit of ivabradine treatment in postural orthostatic tachycardia syndrome (POTS) in participants with Long haul Covid.
  Arms: Ivabradine RCT Arms

SUMMARY:
The purpose of the study is three-fold. The primary aim is to identify the proportion of Long-Haul COVID (LHC) and non-LHC volunteers with relevant symptoms actually have postural orthostatic tachycardia syndrome (POTS). The second is to determine benefit of ivabradine treatment. Ivabradine is a drug approved to treat tachycardia in persons with heart failure. The third is to characterize risk factors and outcomes among volunteers with and without LHC. This will include comparison with COVID-19-positive individuals who did not develop long-COVID symptoms.

The study will improve basic and applied knowledge of LHC and its associated cardiovascular and autonomic consequences. Cellular and molecular characterization of LHC and non-LHC participants will be performed with a nested clinical trial for Ivabradine responsiveness on reduction of tachycardia. It is hoped that a greater understanding of LHC, and related autonomic dysfunction in particular will help to identify treatment paradigms and therapeutic targets for improving recovery and enhancing health for those affected.

DETAILED DESCRIPTION:
The study will first attempt to address the frequency of clinically confirmed POTS in those with persistent COVID-19 symptoms, particularly those symptoms suggestive of autonomic dysfunction.

Those with confirmed POTS or Inappropriate sinus tachycardia (IST) will be randomized to ivabradine or placebo to determine efficacy in reducing heart rate as a putative surrogate for POTS disease as well as effects on POTS symptoms. The biopsychosocial mechanisms of LHC and POTS will also be explored. Specific objectives will be:

1. To assess the frequency and severity of fatigue, dyspnea, headache, and confusion and other suggestive symptoms among volunteers with and without LHC and measure the occurrence of clinically confirmed POTS or IST-in relation to these symptoms.
2. To assess whether treatment with ivabradine will significantly reduce heart rate and improve symptoms and quality of life among subjects manifesting typical POTS or similar autonomic dysregulation.
3. To characterize the immunoinflammatory and genomic factors associated with LHC and POTS among those with LHC. In particular, to determine whether those with POTS have differential expression of genes and/or proteins associated with autonomic nervous system function. To determine whether these factors reflect a genetic predisposition.
4. To determine whether wearable automated ambulatory monitoring with existing FDA-approved devices will permit improved diagnostic accuracy for POTS.
5. To determine the degree to which LHC induced autonomic instability and whether it is associated with induced inflammation and/or dysregulation
6. To evaluate potential contribution of psychological symptoms and the interplay between psychosocial symptoms, quality of life, cognitive symptoms, and physiologic responses induced by LHC.
7. To determine whether LHC improves following vaccination (in the limited number of cases where late vaccination occurs) and/or "breakthrough" clinical COVID-19 infection.
8. Assess whether individuals with LHC have different antibody and/or cellular immune responses to SARS-CoV-2 antigens compared to infected individuals who did not develop LHC.
9. Assess whether specific plasma protein markers of dysregulated blood coagulation, which were significantly correlated with immunothrombosis in severe COVID-19, persist in individuals with LHC.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80
2. History of documented COVID-19 infection of any severity to include a positive COVID-19 PCR, or antibody test
3. Meets criteria for 'long-haul' COVID-19 with symptoms >12 weeks following acute illness
4. Able and willing to provide informed consent and participate for study duration
5. Willing to participate in the nested randomized controlled trial of ivabradine if RCT enrollment criteria are met
6. Access to a primary healthcare provider and proof of health insurance

Inclusion Criteria for non-LHC Cohort

1. Age 18-80
2. History of documented COVID-19 infection of any severity to include a positive COVID-19 PCR, or antibody test
3. Does not meet criteria for 'long-haul' COVID-19
4. Able and willing to provide informed consent and participate for study duration
5. Willing to participate in the nested randomized controlled trial of ivabradine if RCT enrollment criteria are met
6. Access to a primary healthcare provider and proof of health insurance

Inclusion Criteria for POTS RCT:

1. Age 18-80; Meets criteria for 'long-haul' COVID-19

   1. Documented history of COVID-19 infection made available to study team 1914
   2. Lack of documented history, but evidence of infection from sensitive antibody tests
2. Able and willing to provide informed consent and participate for study duration
3. Volunteers with or without LHC combined with POTS based on an increase in comparing the supine heart rate to standing heart rate >20 beats per minute with a drop in systolic blood pressure less than 20 mm Hg or a drop in diastolic blood pressure less than 10 mm Hg will be included, OR additionally, volunteers with or without LHC and a 24-hour mean heart rate of 90 beats per minute or more (in sinus rhythm) will be diagnosed with IST and be included.
4. For females of childbearing age - willing to use a highly effective form of contraceptive with <1% failure rate or practice abstinence for the duration of the study

Exclusion Criteria:

1. Resting heart rate <60 bpm
2. Atrial fibrillation
3. Supraventricular tachycardia
4. Allergic reaction or known contraindications to study drug

   1. Acute decompensated heart failure
   2. Clinically significant hypotension, defined as a drop in systolic BP >20 mmHg or drop in diastolic >10 mmHg during orthostatic vital signs testing.
   3. Sick sinus syndrome, sinoatrial block or 3rd degree AV block, unless a functioning demand pacemaker is present
   4. Clinically significant bradycardia
   5. Severe hepatic impairment
   6. Pacemaker dependence (heart rate maintained exclusively by the pacemaker)
   7. Concomitant use of cytochrome P450 3A4 (CYP3A4) inhibitors or inducers
5. Pregnant/lactating females
6. Impaired gastrointestinal absorption that would preclude oral drug administration
7. Taking any of the following without discontinuation in consultation with the volunteer's healthcare provider and a one-week washout period:

   1. ivabradine
   2. beta-blockers
   3. calcium- channel blockers
   4. cholinesterase inhibitors (pyridostigmine),
   5. vasoconstrictors (midodrine, octreotide, droxidopa, stimulants)
   6. sympatholytics (clonidine, methyldopa)
   7. blood volume enhancers (fludrocortisone, desmopressin, salt supplementation)
   8. oral ketoconazole (contraindicated)
8. Acute suicidality identified at screening

   -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in standing heart rate following 3 months treatment. | 3 months
  The primary endpoint will be a reduction in standing heart rate at 3 months. Up to 200 evaluable subjects will be enrolled in the general LHC cohort with the expectation that at least 20% of those recruited will have POTS or otherwise IST causing symptoms appropriate for enrollment to the nested RCT (ivabradine vs. placebo). This will yield an RCT study population of at least 40 evaluable subjects. Study recruiting will be aimed at volunteers with features of POTS. Drop-outs in all cohorts may be replaced.

CONTACTS AND LOCATIONS:
Overall Officials: David L Saunders, MD, MPH, Principal Investigator — Uniformed Services University of the Health Sciences; Mark C Haigney, MD, FAHA, Study Chair — Uniformed Services University of the Health Sciences
Locations (1):
- Uniformed Services University, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saunders D, Arnold TB, Lavender JM, Bi D, Alcover K, Hellwig LD, Leazer ST, Mohammed R, Markos B, Perera K, Shaw D, Kobi P, Evans M, Mains A, Tanofsky-Kraff M, Goguet E, Mitre E, Pratt KP, Dalgard CL, Haigney MC. Comparative cohort study of post-acute COVID-19 infection with a nested, randomized controlled trial of ivabradine for those with postural orthostatic tachycardia syndrome (the COVIVA study). Front Neurol. 2025 Jul 7;16:1550636. doi: 10.3389/fneur.2025.1550636. eCollection 2025. PMID 40692561

DOCUMENTS (1):
  • Informed Consent Form (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT05481177/ICF_000.pdf